CLINICAL TRIAL: NCT04798118
Title: A Study on Toilet Bronchoscopy In Respiratory ICU, Assiut University Hospital
Brief Title: Role of Toilet Bronchoscopy in RICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaimaa Ali Mohammed, Assistant lecturer,chest department and tuberculosis, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Toilet Bronchoscope
Record Dates: First submitted 2021-03-08; First posted 2021-03-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2022-08

CONDITIONS: COPD; Asthma; Cystic Fibrosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group treated with toilet bronchoscope (Experimental): Toilet bronchoscopy will be done as supportive care to sixty five (COPD,asthma,cystic bronchiectasis ) mechanically ventilated patients who fulfill the following criteria :
  1. Copious secretion
  2. Radiologically diagnosed atelectasis and absent air-bronchograms. Standard care of treatment will be carried out then assessment of a radiological, gasometric improvement and lung mechanics changes.
  Interventions: Procedure: toilet bronchoscope
- group treated with standered care (Active Comparator): sixty five (COPD,asthma,cystic bronchiectasis ) mechanically ventilated patients who fulfill the following criteria :
  1. Copious secretion
  2. Radiologically diagnosed atelectasis and absent air-bronchograms. Standard care of treatment will be carried out then assessment of a radiological, gasometric improvement and lung mechanics changes.
  Interventions: Procedure: toilet bronchoscope

INTERVENTIONS:
Procedure: toilet bronchoscope — Toilet bronchoscopy will be done by infuse normal saline or N-Acetylcysteine with a syringe, observing the flow of saline at the distal tip of the bronchoscope then suction intra bronchial visible secretions during the procedure and also suction of specific lobe guided by radiological finding in the patient A chest X-ray will be routinely performed prior and after the procedure, HRCT is mandatory when chest x-ray not clearly defining the collapse monitoring of heart rate, oxygen saturation, ventilator parameters, and arterial blood pressure will be done

SUMMARY:
Toilet bronchoscopy is a potentially therapeutic intervention to aspirate retained secretions within the endotracheal tube and airways and revert atelectasis. Aspiration of airway secretions is the most common indication to perform a therapeutic bronchoscopy in the intensive care unit (ICU) .

Toilet bronchoscopy is particularly beneficial when retained secretions are visible during the procedure and when air-bronchograms are not present at the chest radiograph. It is also beneficial when there is an indication to reverse lobar atelectasis, rather than simply to remove accumulated mucus.

Toilet bronchoscopy is used in lobar and complete lung collapse in mechanically ventilated patients who fail to respond to treatments such as physiotherapy or recruitment manoeuvres.

The success rates (defined as radiographic improvement on chest X-ray [CXR] or an improved PaO2/PAO2 ratio) in the ICU patient population had.

Patients with acute hypoxaemic respiratory failure may already be on non-invasive ventilation (NIV), or require NIV preemptively for Fiberoptic Bronchoscopy (FB). These patients should be considered high risk for requiring intubation post-procedure; therefore, Fiberoptic Bronchoscopy should be performed by an experienced operator in a setting allowing facilities to safely secure the airways. NIV with early therapeutic FB rather than mechanical ventilation can help avoid intubation and reduce tracheostomy rate. Hospital mortality, duration of ventilation, and hospital stay remain similar

DETAILED DESCRIPTION:
Aim Of Work To study the value of toilet bronchoscopy in

1. Mechanical ventilated patients with chest disease and copious secretion.
2. Mechanical ventilated patients diagnosed to have atelectasis radiologically.
3. Patients on non-invasive ventilation with chest diseases and copious secretion
4. Compare Different types of mucolytics during toilet bronchoscopy in mechanically ventilated patients.
5. Compare Different types of sedations during toilet bronchoscopy in mechanically ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* • Patients on mechanical ventilation with underlying dieases that are characterized with mucus overproduction such as asthma, chronic obstructive pulmonary disease (COPD), bronchiectasis, and cystic fibrosis.

  * Patients on mechanical ventilation with visible large amount of sputum during suction in order to clear secretions.
  * Patients on mechanical ventilation with radiologically diagnosed atelectasis and absent air-bronchograms
  * Patient on NIV who was benefit from toilet bronchoscopy to clear retained secretion.

Exclusion Criteria:Absolute contraindications

* Absence of consent from the patient or his/her representative.
* Inability to adequately oxygenate the patient during the procedure.
* Current myocardial ischaemia.
* Significant haemodynamic instability.
* Life-threatening cardiac arrhythmias.
* Current significant bronchospasm.
* Undrained pneumothorax.

Relative contraindications

* Thrombocytopenia (platelet count ≤50,000 platelets/mm).
* INR of 2 or greater, or an elevated PTT.
* BUN >30.
* severe tracheal obstruction.
* Recent myocardial ischaemia and/or unstable angina.
* Intracranial hypertension.
* Poorly-controlled heart failure.
* Recent oral intake.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
1- percent of patients develop radiological improvement | 12 months
  assessed improvement of atelectasis by chest x-ray or HRCT
2- improvement of hypoxemia | 12months
  assessed by sao2/fio2 or pao2/fio2 before and after procedure
3-Lung mechanics reduction post procedure in mechanical ventilated patients | 12 months
  resistance measured by cm H2o /Liter/ second
Lung mechanics improvement post procedure in mechanical ventilated patients | 12 months
  assessed by static compliance measured by ml/cm H2o

SECONDARY OUTCOMES:
length of ICU stay | 12 months
  measured by days
length of hospital stay | 12 months
  measured by days
occurrence of complications | 12 months
  developed or not
4-Hospital mortality | 12 months
  percent in each group

CONTACTS AND LOCATIONS:
Overall Officials: Saher f youssif, Principal Investigator — Assiut University
Locations (1):
- Assuit university hospital, Asyut, Egypt

REFERENCES:
- [Background] Marini JJ, Pierson DJ, Hudson LD. Acute lobar atelectasis: a prospective comparison of fiberoptic bronchoscopy and respiratory therapy. Am Rev Respir Dis. 1979 Jun;119(6):971-8. doi: 10.1164/arrd.1979.119.6.971. PMID 453712
- [Background] Snow N, Lucas AE. Bronchoscopy in the critically ill surgical patient. Am Surg. 1984 Aug;50(8):441-5. PMID 6465691
- [Background] Kreider ME, Lipson DA. Bronchoscopy for atelectasis in the ICU: a case report and review of the literature. Chest. 2003 Jul;124(1):344-50. doi: 10.1378/chest.124.1.344. PMID 12853543
- [Background] Jelic S, Cunningham JA, Factor P. Clinical review: airway hygiene in the intensive care unit. Crit Care. 2008;12(2):209. doi: 10.1186/cc6830. Epub 2008 Mar 31. PMID 18423061
- [Background] Jose RJ, Shaefi S, Navani N. Sedation for flexible bronchoscopy: current and emerging evidence. Eur Respir Rev. 2013 Jun 1;22(128):106-16. doi: 10.1183/09059180.00006412. PMID 23728864